CLINICAL TRIAL: NCT05025241
Title: An Open-Label Study of the Safety, Tolerability, and Pharmacokinetics of Oral NNZ-2591 in Phelan-McDermid Syndrome (PMS-001)
Brief Title: An Open-Label Study of Oral NNZ-2591 in Phelan-McDermid Syndrome (PMS-001)
Acronym: PMS-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-2591-PMS-001
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Phelan-McDermid Syndrome
Keywords: Phelan-McDermid Syndrome
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome | interventions — cyclo-L-glycyl-L-2-allylproline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNZ-2591 (Experimental): NNZ-2591 oral solution (50mg/mL) to be administered twice daily dose for 13 weeks.
  Interventions: Drug: NNZ-2591

INTERVENTIONS:
Drug: NNZ-2591 — NNZ-2591 oral solution (50mg/mL) to be administered twice daily dose for 13 weeks.
  Other Names: Cyclo-L-Glycyl-L-2-Allylproline

SUMMARY:
A study of the safety, tolerability and pharmacokinetics of NNZ-2591 and measures of efficacy in children and adolescents with Phelan-McDermid Syndrome.

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate the safety, tolerability and pharmacokinetics of treatment with NNZ-2591 oral solution in children and adolescents with Phelan-McDermid Syndrome. The secondary purpose is to investigate measures of efficacy. Subjects will receive treatment with NNZ-2591 oral solution (50 mg/mL) doses for a total of 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of PMS with a documented disease-causing genetic abnormality of SHANK3.
2. Males or females aged 3-12 years.
3. Body weight of 12 kg or higher at Screening.
4. Subjects with a Clinical Global Impression - Severity (CGI-S) score of 4 or greater at the Screening visit.
5. Not actively undergoing regression or loss of skills, defined as no persistent loss of previously acquired developmental skills for a period within 3 months of the Screening visit
6. Each subject must be able to swallow the study medication provided as a liquid solution.
7. Caregiver(s) must have sufficient English language skills.

Exclusion Criteria:

1. Body weight < 12kg at screening
2. Clinically significant abnormalities in safety laboratory tests and vital signs at Screening.
3. Abnormal QTcF interval or prolongation at Screening.
4. Any other clinically significant finding on ECG at the Screening visit.
5. Positive for severe acute respiratory syndrome coronavirus 2 (SARSCoV- 2) and previous COVID 19 infection with last 12 months that required hospitalization
6. Unstable or changes Psychotropic treatment 2 weeks prior to screening .
7. Excluded concomitant treatments.
8. Actively undergoing regression or loss of skills.
9. Unstable seizure profile.
10. Current clinically significant renal conditions and abnormalities
11. Current clinically significant cardiovascular, renal, hepatic, gastrointestinal, respiratory, endocrine disease, or clinically significant organ impairment.
12. Current clinically significant hypo or hyperthyroidism, Type 1 or Type 2 diabetes mellitus requiring insulin (whether well controlled or uncontrolled), or uncontrolled Type 1 or Type 2 diabetes.
13. Has planned surgery during the study.
14. History of, or current, cerebrovascular disease or brain trauma.
15. History of, or current catatonia or catatonia-like symptoms.
16. History of, or current, malignancy.
17. Current major or persistent depressive disorder (including bipolar depression).
18. Significant, uncorrected visual or uncorrected hearing impairment.
19. Allergy to strawberry.
20. Positive pregnancy test
21. Subject is judged by the Investigator or Medical Monitor to be inappropriate for the study

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Shaw, Study Director — Neuren Pharmaceuticals
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neumeyer AM, Srivastava S, Holder JL, Milad MA, Squires L, Jones NE, Glass L, Berry-Kravis E. NNZ-2591 in Children and Adolescents With Phelan-McDermid Syndrome: Single-Group, Open-Label, Phase 2 Trial Results. Neurol Genet. 2025 Dec 23;12(1):e200338. doi: 10.1212/NXG.0000000000200338. eCollection 2026 Feb. PMID 41450730

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 4 academic medical centers between August 2022 and June 2023. The first participant entered screening on 08 August 2022, and the last participant entered screening on 22 June 2023. Of 23 consented participants, 18 met eligibility criteria and were enrolled into the study. Enrolled participants received NNZ2591 12 mg/kg by liquid oral dose twice daily
Pre-assignment Details: Following consent, participants underwent 4 weeks of screening for eligibility. If successful, participants were enrolled and commenced open-label active treatment.
Groups:
- NNZ-2591: All enrolled participants
Period: Screening
Arm/Group | NNZ-2591
Started | 23
Completed | 18
Not Completed | 5
Not completed — Failed Screening | 5
Period: Treatment and Follow Up
Arm/Group | NNZ-2591
Started | 18
Completed | 15
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Intention to treat
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : White | 16
  Race : Black or African American | 1
  Race : Asian | 0
  Race : Native Hawaiian or other Pacific Islander | 0
  Race : American Indian or Alaska Native | 0
  Race : Multi Racial | 1
  Race : Other | 0
  Ethnicity : Hispanic or Latino | 3
  Ethnicity : Not Hispanic or Latino | 15
Height (cm) [Mean (Standard Deviation); unit: cm] | 130.6 (15.15)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 30.4 (10.75)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 17.4 (3.48)
PMS Genotype [Count of Participants; unit: Participants]
  Terminal Deletion - Class I | 7
  Terminal Deletion - Class II | 3
  Ring 22 | 0
  Unbalanced Translocation | 0
  Interstitial Deletion | 1
  SHANK 3 variant/mutation | 6
  Other | 1
History of regression [Count of Participants; unit: Participants]
  Yes | 11
  No | 7
Autism Mental Status Exam [Mean (Standard Deviation); unit: score on a scale] — The AMSE is an observational assessment that looks at 8 items of social, communicative and behavioral functioning in individuals with Autism Spectrum Disorder, with each item yielding a potential score of 0, 1 or 2, with range of 0-16. Higher scores indicate greater levels of impairment.
  score on a scale | 7.8 (2.05)
Seizure Types [Count of Participants; unit: Participants] — Population: Only 2 participants recorded seizures at enrollment
  Participants
    Simple Partial: number analyzed (Participants) | 2
    Simple Partial | 0
    Complex Partial: number analyzed (Participants) | 2
    Complex Partial | 1
    Atonic: number analyzed (Participants) | 2
    Atonic | 1
    Tonic: number analyzed (Participants) | 2
    Tonic | 1
    Clonic: number analyzed (Participants) | 2
    Clonic | 0
    Tonic-Clonic: number analyzed (Participants) | 2
    Tonic-Clonic | 1
    Myoclonic: number analyzed (Participants) | 2
    Myoclonic | 0
    Absence/Atypical Absence: number analyzed (Participants) | 2
    Absence/Atypical Absence | 0
    Not Actual Seizure/Spells: number analyzed (Participants) | 2
    Not Actual Seizure/Spells | 0
    Other: number analyzed (Participants) | 2
    Other | 1
Seizure Characteristics at baseline [Number; unit: participants]
  Change in awareness | 2
  Loss of urine or bowel control | 0
  Loss of ability to communicate | 2
  Automatic repeated movements | 0
  Rhythmic jerking muscle | 2
  Falls if sitting or standing | 0
  Head drops | 1
  Warning before seizure occurred | 0
  Common triggers | 0
  Muscle stiffness | 1
  Muscle twitch | 1
  Other | 1
Stanford-Binet Intelligence Scale (NVIQ) Standard Score [Mean (Standard Deviation); unit: score on a scale] — The Stanford Binet Non Verbal IQ (NVIQ) is a normed combined score taken from the 5 non verbal subtests. The score represents an individuals performance on the 5 nonverbal subtests of the exam with a range of 40-160, with higher scores indicating greater non verbal intelligence. Population: Participants who could not be assessed on the Stanford-Binet Intelligence (SB-5) due to their developmental level were assessed using the Mullen Scales of Early Learning instead.
  score on a scale
    number analyzed (Participants) | 9
    (all) | 47.7 (5.39)
Stanford-Binet Intelligence Scale (NVIQ) z deviation score [Mean (Standard Deviation); unit: score on a scale] — The z deviation score measures how far an individual's performance deviates from the mean performance of the normative sample on a specific subtest or composite score.
  Formula:
  Z = (X-μ)/σ
  Where:
  Z: The z-score (z deviation score). X: The individual's raw or scaled score. μ: The mean score of the normative sample. σ: The standard deviation of the scores in the normative sample.
  A positive z-score indicates a score above the mean. A negative z-score indicates a score below the mean. Population: Participants who could not be assessed on the Stanford-Binet Intelligence (SB-5) due to their developmental level were assessed using the Mullen Scales of Early Learning instead.
  score on a scale
    number analyzed (Participants) | 9
    (all) | 40.9 (17.2)
Mullen Scales of Early Learning Non-Verbal Developmental Quotient Score [Mean (Standard Deviation); unit: score on a scale] — The Non-Verbal Developmental Quotient (NVDQ) on the Mullen Scales of Early Learning assesses a child's non-verbal cognitive abilities by combining t-scores from the two non-verbal subscales scores of the Mullen Scales:
  1. Visual Reception (VR) subscale
  2. Fine Motor (FM) subscale
  3. This effectively rescales the score back to a quotient scale similar to an IQ score, where the mean is 100 and the standard deviation is 15.
  5 Scores > 100 indicate higher non-verbal developmental abilities, while scores < 100 suggest potential delays. Population: Includes only participants who were unable to be assessed on the Stanford-Binet Intelligence (SB-5) due to their developmental level.
  score on a scale
    number analyzed (Participants) | 8
    (all) | 15.7 (7.25)
Presence of co-morbid psychiatric disorders [Number; unit: participants]
  Autism Spectrum Disorder (ASD) | 14
  BiPolar Disorders | 0
  Attention Deficit Disorder | 5
  Obsessive Compulsive Disorder | 0
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: To examine the incidence, severity and frequency of adverse events (AEs), including serious adverse events (SAEs) during treatment with NNZ-2591.
Time Frame: 13 weeks
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
Participants
  Participants with any AE | 17
  Participants with TEAE | 17
  Participants with Serious TEAE | 1
  Participants who discontinued due to TEAE | 3
  Participants with mild TEAE | 11
  Participants with moderate TEAE | 5
  Participants with severe TEAE | 1

2. Primary Outcome: Pharmacokinetic - Mean AUC24
Description: Approximately nine sparse pharmacokinetic (PK) samples were collected from each participant under steady-state conditions. These samples were taken at pre-dose, 1-3 hours post-dose, and/or 4-7 hours post-dose during Weeks 2, 6, and 13. The individual pharmacokinetic parameters for NNZ-2591, including half-life (t1/2) and area under the curve over 24 hours (AUC24), were derived using subject-level concentration-time profiles from the study population model.
Time Frame: Pre-dose, 1-3 h post-dose and/or 4-7 h post-dose at Weeks 2, 6 and 13.
Population: PK Population
Measure: Mean (Standard Deviation); unit: µg.h/mL
Groups:
- PK Population: All participants enrolled in this study who receive the study drug through to the morning dose of Week 2 (Visit 5) as a minimum, and who undergo PK sample collection at least one of the specified post-dose time point(s).
Arm/Group | PK Population
Number analyzed (Participants) | 18
µg.h/mL | 411 (116)

3. Primary Outcome: Pharmacokinetic - t1/2
Description: as for outcome 2
Time Frame: Pre-dose, 1-3 h post-dose and/or 4-7 h post-dose at Weeks 2, 6 and 13.
Population: All participants enrolled in this study who receive the study drug through to the morning dose of Week 2 (Visit 5) as a minimum, and who undergo PK sample collection at least one of the specified post-dose time point(s).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PK Population
Number analyzed (Participants) | 18
hours | 8.02 (2.33)

4. Secondary Outcome: CGI-I
Description: Phelan-McDermid Syndrome-specific Clinical Global Impression of Improvement Scale (CGI-I) - Overall Improvement Score on a 7 point Likert scale (1-7) where lower scores are better.
Time Frame: CGI-I was assessed at Weeks 6, 13/EOT & 15. Overall improvement scores relate to Week 13/EOT visit.
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | 2.4 (0.86)
Statistical Analysis 1: Comparison: NNZ-2591; Efficacy endpoints were analyzed using a Wilcoxon signed rank test on the paired participant data from baseline to EOT (Visit 16), when applicable. Baseline values were based on the average non-missing values of visits 1, 2, and 3 for assessments collected at more than one visit during the Screening/Baseline period. Descriptive statistics were used to summarize the data. For total scores, waterfall plots, and histograms were created at the EOT visit with plots for all participants; Test type: Other; p < 0.0001, Wilcoxon Signed rank

5. Secondary Outcome: CIC
Description: Caregiver Impression of Improvement: Measured on a 7 point Likert scale (1-7) where lower scores are better.
Time Frame: CIC was assessed at Week13/EOT
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | 2.7 (1.02)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0003, Wilcoxon Signed rank

6. Secondary Outcome: CGI-S
Description: Phelan-McDermid syndrome-specific Clinical Global Impression Scale-Severity (CGI-S) -Change from baseline on Overall Score. Based on a 7 point Likert scale (1-7) where a lower score is better.
Time Frame: Change in score assessed from baseline (visit 3, week 0) to visit 16 (week 13/EOT).
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | -0.4 (0.5)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — Change from baseline; p = 0.0156, Wilcoxon Signed rank

7. Secondary Outcome: Top 3 Concerns
Description: Caregiver Top 3 Concerns - Total Concerns Severity: Change from baseline. The range of scores was (0-30) for total concerns, with higher scores being worse
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in overall improvement score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | -5.9 (5.86)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — Change from baseline; p = 0.0005, Wilcoxon Signed rank

8. Secondary Outcome: MB-CDI
Description: MacArthur-Bates Communicative Development Inventory (MB-CDI) - change from baseline. Range of scores was (0-792) with higher scores being better.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16).
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | 12.3 (35.19)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0647, Wilcoxon Signed rank

9. Secondary Outcome: ORCA
Description: Observer-Reported Communication Ability (ORCA) - Change from baseline in Total Score. Range of Scores was (25.8-83.8) with higher scores being better
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in Total Score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | 1.9 (4.22)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — Change from baseline; p = 0.0984, Wilcoxon Signed rank

10. Secondary Outcome: ABC-2
Description: Aberrant Behavior Checklist-2 (ABC-2) - Total score: Change from baseline. Range of scores was (0-174) with higher scores being worse
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in total score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | -17.2 (19.65)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — Change from baseline; p = 0.0013, Wilcoxon Signed rank

11. Secondary Outcome: CSHQ
Description: Child Sleep Habits Questionnaire (CSHQ) - Change from baseline in Total Score. Range of scores was (33-99) with higher scores being worse.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in total score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | -3.6 (5.68)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — Change from baseline; p = 0.0191, Wilcoxon Signed rank

12. Secondary Outcome: GIHQ
Description: Gastrointestinal Health Questionnaire (GIHQ) - Total Frequency Score: Change from Baseline. Range of scores was (0-212) with higher scores being worse.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in total frequency score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | -9.6 (10.8)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — change from baseline; p = 0.0013, Wilcoxon Signed rank

13. Secondary Outcome: VABS-3
Description: Vineland Adaptive Behavior Scales-3, Change from baseline in Composite Standard Score. Range of scores was (20-140) with higher scores being better.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in composite standard score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | 2.8 (7.82)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — change from baseline; p = 0.1710, Wilcoxon Signed rank

14. Secondary Outcome: QL-Disability
Description: Quality of Life Inventory-Disability (QL-Disability) Overall Score - change from baseline. Range of scores was (0-100) with higher scores being better.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in overall score score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | 6.1 (8.91)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — change from baseline; p = 0.0066, Wilcoxon Signed rank

15. Secondary Outcome: ICND
Description: Impact of Childhood Neurological Disability (ICND) - Change from baseline in overall quality of life rating. Range of (1- 6) for quality of life rating, with higher scores indicating greater impact.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in overall quality of life rating score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | 0.3 (0.69)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — change form baseline; p = 0.1094, Wilcoxon Signed rank

16. Secondary Outcome: PMS-DSRS
Description: PMS Clinician Domain Specific Rating Scale - Change from baseline in overall severity score. Range of Scores Was (0-20) With Higher Scores Being Worse.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in overall severity score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | -0.9 (1.69)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — change from baseline; p = 0.0156, Wilcoxon Signed rank

17. Secondary Outcome: Behavior Problems Inventory - Short Form
Description: Total Frequency Score - Change from Baseline. Range of scores was (0-4) for each of 30 behaviors, total range (0-120), with lower scores being better.
Time Frame: Change from baseline (visit 3, week 0) to visit 13/EOT (week 16) in total frequency score.
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNZ-2591
Number analyzed (Participants) | 18
score on a scale | -5.1 (9.41)
Statistical Analysis 1: Comparison: NNZ-2591; [analysis description as in outcome 4, analysis 1]; Test type: Other — change from baseline; p = 0.0326, Wilcoxon Signed rank

ADVERSE EVENTS:
Time Frame: 15 weeks for each participant starting on date of first dose
Description: Once eligibility was confirmed, subjects were dosed at a starting dose of 4 mg/kg twice daily (BID). Doses were titrated to 8 mg/kg at week 2 and to 12 mg/kg at week 6. The mg/kg dosing was based on the subject's weight at baseline. Subjects received treatment with NNZ-2591 for a total of 13 weeks.
Arm/Group | NNZ-2591
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNZ-2591 (N=18)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNZ-2591 (N=18)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Pyrexia (General disorders) | 3 (3)
Covid 19 (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2)
Otitis Media (Infections and infestations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Psychomotor Hyperactivity (Nervous system disorders) | 4 (4)
Somnolence (Nervous system disorders) | 3 (3)
Aggression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT05025241/Prot_003.pdf
  • Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT05025241/SAP_004.pdf